CLINICAL TRIAL: NCT02834819
Title: A Randomized Controlled Trial of Nebulized 3% Hypertonic Saline vs. Standard of Care in Patients With Bronchiolitis
Brief Title: Nebulized 3% Hypertonic Saline vs. Standard of Care in Patients With Bronchiolitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-0092
Record Dates: First submitted 2016-04-01; First posted 2016-07-15 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; hypoxia; hypertonic saline
MeSH Terms: conditions — Bronchiolitis; Hypoxia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypertonic Saline (Experimental): Patients randomized to the hypertonic saline group will be administered one nebulized treatment of 3% hypertonic saline. They will also receive what is considered standard of care, which includes suctioning and supportive care as needed.
  Interventions: Drug: 3% Nebulized Hypertonic Saline
- No treatment (No Intervention): Patients in the "No treatment" arm will receive no additional treatment other than standard of care, which includes suctioning and supportive care as needed.

INTERVENTIONS:
Drug: 3% Nebulized Hypertonic Saline
  Arms: Hypertonic Saline

SUMMARY:
The purpose of this study is to determine whether nebulized 3% hypertonic saline is more effective than the current standard of care in the treatment of viral bronchiolitis in children.

DETAILED DESCRIPTION:
This will be a prospective, randomized controlled single-blinded study of patients 3-18 months of age presenting to the Children's Hospital Colorado ED during bronchiolitis season, diagnosed with mild to moderate bronchiolitis and persistent hypoxia and started on the Children's Hospital Colorado Home Oxygen pathway (see attached clinical care guideline). Investigators aim to enroll 220 patients. Patients will be identified by research assistants in the ED, based on physician diagnosis of bronchiolitis, with hypoxia requiring < 0.5L oxygen by NC. A research assistant will approach the family and go through the informed consent process. If consent is obtained, the patient will then be randomized to one of the two study arms via a computer generated randomization table. In order to arrange for respiratory therapy, the research assistants will not be blinded. There will be an age block randomization scheme, and therefore patients aged 3-12 months will be randomized separately from patients 12.1-18 months to ensure equal distribution of age ranges in each arm.

The experimental arm will consist of patients who receive a nebulized treatment of 4ml of 3% hypertonic saline, administered by a respiratory therapist, as well as supportive care as needed. Patients in the control arm will receive supportive care only, the current standard of care at Children's Hospital Colorado. The pharmacist will randomize patients as noted above. After consent is obtained the provider will perform a pre-intervention clinical severity score evaluation to patients in both study arms utilizing the clinical severity score tool described by Wang et al.19 Respiratory therapy will then provide the nebulized treatment for those patients randomized to receive hypertonic saline. Removal of equipment following treatment will aid in ensuring blinding of physicians to treatment arm. At 90 minutes after treatment with hypertonic saline or after the order is placed for patients in the control arm, patients in both arms will undergo a second clinical severity score by the provider. At that time the provider will turn off the oxygen administered to both treatment arms for a room air challenge. The RN will be notified that the patients are off oxygen therapy and will restart oxygen if patient has saturations < 87% (as indicated by continuous pulse oximetry) and oxygen will be restarted at 0.5L by NC.

Patients in both arms who are no longer requiring oxygen will be observed for a minimum of 4 hours to ensure they remain stable on room air, have appropriate oral intake, and sleep without de-saturation. At any point if a patient who was weaned off oxygen becomes hypoxic (saturations < 87%), requiring < 0.5L oxygen NC they will return to the home oxygen observation protocol. If during this period of observation any patient requires > 0.5L oxygen during wake or sleep periods, is not taking adequate oral intake, demonstrates respiratory distress, or at physician discretion, patient may be admitted to the inpatient service for further management.

Patients in both arms will receive follow-up phone calls to assess duration and amount of oxygen, as well as adverse outcomes. Patients discharged home on room air will receive 1 phone call on post-discharge day #7 (range 6-8). Patients discharged home on oxygen will receive a phone call on day #7 (range 6-8). Calls will be made for the study by the study investigators or by the Emergency Department (ED) research assistants. During the follow-up phone call, caregivers will be asked about Primary Care Physician (PCP) follow-up visits, any future scheduled PCP visits, any adverse events including increased work of breathing, increased oxygen requirement, repeat ED visits to researchers or other institutions, outside hospital admissions, intensive care unit admission or intubations, and any instructions for weaning oxygen given by PCP. If parents have questions or concerns, these questions will be directed to a nurse, fellow, or attending provider.

Data from each subject will be collected on a data collection sheet for the follow-up phone call and PCP call. Data will then be entered into a database on a secure server and de-identified. All identifiers will be removed from the data set.

The Electronic Health Record will be reviewed to verify return visits. If return visits are documented in EPIC (electronic health records software), data on type of admission (general pediatrics or intensive care unit) and any advanced airway intervention such as intubation, continuous positive airway pressure (CPAP).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Children's Hospital Colorado ED
* ≥3 to ≤18 months of age
* Diagnosed with bronchiolitis
* Have persistent hypoxia following initial supportive care measures as outlined by Children's Hospital Colorado Bronchiolitis Clinical Care Guideline
* Started on Children's Hospital Colorado Home Oxygen Pathway

Exclusion Criteria:

* Patients who do not qualify for the Clinical Care Guideline for Home oxygen for Bronchiolitis
* Previous history of wheezing
* History of reactive airway disease
* History of underlying heart disease
* Require >0.5L oxygen

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cortney Braund, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zorc JJ, Hall CB. Bronchiolitis: recent evidence on diagnosis and management. Pediatrics. 2010 Feb;125(2):342-9. doi: 10.1542/peds.2009-2092. Epub 2010 Jan 25. PMID 20100768
- [Background] American Academy of Pediatrics Subcommittee on Diagnosis and Management of Bronchiolitis. Diagnosis and management of bronchiolitis. Pediatrics. 2006 Oct;118(4):1774-93. doi: 10.1542/peds.2006-2223. PMID 17015575
- [Background] Yorita KL, Holman RC, Sejvar JJ, Steiner CA, Schonberger LB. Infectious disease hospitalizations among infants in the United States. Pediatrics. 2008 Feb;121(2):244-52. doi: 10.1542/peds.2007-1392. PMID 18245414
- [Background] Kini NM, Robbins JM, Kirschbaum MS, Frisbee SJ, Kotagal UR; Child Health Accountability Initiative. Inpatient care for uncomplicated bronchiolitis: comparison with Milliman and Robertson guidelines. Arch Pediatr Adolesc Med. 2001 Dec;155(12):1323-7. doi: 10.1001/archpedi.155.12.1323. PMID 11732950
- [Background] Pelletier AJ, Mansbach JM, Camargo CA Jr. Direct medical costs of bronchiolitis hospitalizations in the United States. Pediatrics. 2006 Dec;118(6):2418-23. doi: 10.1542/peds.2006-1193. PMID 17142527
- [Background] Mallory MD, Shay DK, Garrett J, Bordley WC. Bronchiolitis management preferences and the influence of pulse oximetry and respiratory rate on the decision to admit. Pediatrics. 2003 Jan;111(1):e45-51. doi: 10.1542/peds.111.1.e45. PMID 12509594
- [Background] Zhang L, Mendoza-Sassi RA, Wainwright C, Klassen TP. Nebulized hypertonic saline solution for acute bronchiolitis in infants. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006458. doi: 10.1002/14651858.CD006458.pub2. PMID 18843717
- [Background] Mai XM, Nilsson L, Kjellman NI, Bjorksten B. Hypertonic saline challenge tests in the diagnosis of bronchial hyperresponsiveness and asthma in children. Pediatr Allergy Immunol. 2002 Oct;13(5):361-7. doi: 10.1034/j.1399-3038.2002.01011.x. PMID 12431196
- [Background] Wark P, McDonald VM. Nebulised hypertonic saline for cystic fibrosis. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD001506. doi: 10.1002/14651858.CD001506.pub3. PMID 19370568
- [Background] Ralston S, Hill V, Martinez M. Nebulized hypertonic saline without adjunctive bronchodilators for children with bronchiolitis. Pediatrics. 2010 Sep;126(3):e520-5. doi: 10.1542/peds.2009-3105. Epub 2010 Aug 16. PMID 20713480

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypertonic Saline: Patients randomized to the hypertonic saline group will be administered one nebulized treatment of 3% hypertonic saline. They will also receive what is considered standard of care, which includes suctioning and supportive care as needed.
  3% Nebulized Hypertonic Saline
Period: Overall Study
Arm/Group | Hypertonic Saline | No Treatment
Started | 9 | 9
Completed | 4 | 9
Not Completed | 5 | 0
Not completed — Did not complete 7 day follow up call. | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypertonic Saline | No Treatment | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 202.22 (109.37) | 255.33 (122.43) | 228.77 (115.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Hospitalization Rate
Description: Effect of nebulized 3% hypertonic saline on hospitalization rate in children with bronchiolitis compared to those who receive the current standard of care
Time Frame: At any point during enrollment visit or up to 7 days after enrollment visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline | No Treatment
Number analyzed (Participants) | 9 | 9
Participants | 2 | 1

2. Primary Outcome: Number of Patients With Persistent Hypoxia
Description: To assess the effect of nebulized hypertonic saline on hypoxia in children with bronchiolitis compared to those who receive current standard of care.
Time Frame: At baseline and 90 minutes post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline | No Treatment
Number analyzed (Participants) | 9 | 9
Participants | 9 | 9

3. Primary Outcome: Need for Supplemental Oxygen After Discharge
Description: To assess the effect of nebulized hypertonic saline on supplemental home oxygen requirement in children with bronchiolitis compared to those who receive the current standard of care.
Time Frame: At time of discharge from the hospital through 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline | No Treatment
Number analyzed (Participants) | 9 | 9
Participants | 9 | 9

4. Secondary Outcome: Pre- Intervention Clinical Severity Score
Description: Clinical severity score taken immediately following randomization, and prior to any intervention to assess change in baseline after intervention and compare change in scores, if any, between the two groups. The Scale utilized was the Clinical Severity Score from Wang et al, which measures respiratory distress in young children. The system assigns scores ranging from 0 to 3 for the following categories: respiratory rate, wheezing, retraction, and general condition. These category scores are then summed to come up with the final Clinical Severity Score. Total scores range from 0 to 12, with higher scores indicating greater severity/worse outcomes.
Time Frame: During Enrollment visit following randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypertonic Saline | No Treatment
Number analyzed (Participants) | 9 | 9
score on a scale | 3.8 (1.8) | 2.7 (2.04)

5. Secondary Outcome: Post-intervention Clinical Severity Score
Description: Clinical severity score taken at time 90 minutes in both arms to assess any change in clinical severity score from baseline. The Scale utilized was the Clinical Severity Score from Wang et al, which measures respiratory distress in young children. The system assigns scores ranging from 0 to3 for the following categories: respiratory rate, wheezing, retraction, and general condition. These category scores are then summed to come up with the final Clinical Severity Score. Total scores range from 0 to 12, with higher scores indicating greater severity/worse outcomes.
Time Frame: During enrollment visit - 90 minutes after randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypertonic Saline | No Treatment
Number analyzed (Participants) | 9 | 9
score on a scale | 2.22 (1.48) | 2.22 (2.22)

6. Secondary Outcome: Unscheduled Return ED Visits
Description: Unscheduled visit to ED within 3 days of enrollment visit.
  Patients in each group will be contacted 7 days after the enrollment visit to see if they had any unscheduled return ED visit within 3 days of the enrollment visit.
Time Frame: Called at 7 days post enrollment visit to assess any visit within 3 days of enrollment visit
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline | No Treatment
Number analyzed (Participants) | 9 | 9
Participants | 0 | 0

7. Secondary Outcome: Adverse Outcomes
Description: Respiratory distress, increased oxygen requirement, advanced airway interventions (NIPPV or intubation).
Time Frame: During enrollment visit or within 7 days following enrollment visit
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline | No Treatment
Number analyzed (Participants) | 9 | 9
Participants | 0 | 0

8. Secondary Outcome: Hospital Admission After Discharge
Description: Admission to any hospital institution within 7 days following enrollment visit
Time Frame: Within 7 days following discharge from enrollment visit
Population: 5 patients did not complete the 7 day phone call and were not able to be analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline | No Treatment
Number analyzed (Participants) | 4 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Hypertonic Saline | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No